CLINICAL TRIAL: NCT01688037
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NBI-98854 for the Treatment of Tardive Dyskinesia in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: NBI-98854 for the Treatment of Tardive Dyskinesia in Subjects With Schizophrenia or Schizoaffective Disorder (KINECT Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-1201
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NBI-98854 50 mg (Experimental): NBI-98854 50 mg administered as two (2) 25 mg capsules by mouth, taken every morning between 7:00am - 10:00am for 6 weeks.
  Interventions: Drug: NBI-98854
- NBI-98854 100 mg and 50 mg (Experimental): NBI-98854 100 mg administered as two (2) 50 mg capsules taken every morning between 7:00am - 10:00am for 2 weeks. After 2 weeks, NBI-98854 50 mg administered by two (2) 25 mg capsules by mouth, taken every morning between 7:00am - 10:00am for remaining 4 weeks.
  Interventions: Drug: NBI-98854
- Placebo (Placebo Comparator): Capsule containing no active substance, manufactured to mimic NBI-98854 25 mg and 50 mg capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-98854 — 25 mg capsule
  Arms: NBI-98854 100 mg and 50 mg; NBI-98854 50 mg
Drug: NBI-98854 — 50 mg capsule
  Arms: NBI-98854 100 mg and 50 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of two doses (50 and 100 mg) of NBI-98854 administered once daily for the treatment of Tardive Dyskinesia (TD) symptoms.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy, safety, and tolerability of two doses (50 and 100 mg) of NBI-98854 administered once daily for up to 2 weeks. The study will also allow for an evaluation of the efficacy of NBI-98854 50 mg once daily for up to 6 weeks and the safety and tolerability of NBI 98854 50 mg once daily for up to 12 weeks.

The double-blind placebo-controlled treatment period the study has three arms:

* NBI-98854 50 mg once daily for 6 weeks
* NBI-98854 100 mg once daily for 2 weeks followed by 50 mg once daily for the remaining 4 weeks
* placebo

At the end of the 6-week placebo-controlled double-blind treatment period, subjects will continue in the study for an additional 6-week open-label period where all subjects who have completed the double-blind treatment period will receive NBI-98854 50 mg once daily. Two and four weeks after the last dose of study drug, follow-up assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of schizophrenia or schizoaffective disorder and a clinical diagnosis of neuroleptic-induced tardive dyskinesia for at least 3 months prior to screening.
* Be receiving a stable dose of antipsychotic medication for a minimum of 30 days before study start. Subjects who are not using antipsychotic medication must have stable psychiatric status.
* Have the doses of concurrent medications and the conditions being treated be stable for a minimum of 30 days before study start and be expected to remain stable during the study.
* Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal birth control during the study.
* Female subjects must not be pregnant.
* Be in good general health and expected to complete the clinical study as designed.
* Have a body mass index (BMI) of 18 to 38 kg/m2 (both inclusive).
* Have a negative urine drug screen (negative for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids) at screening and study start, except for any subject receiving a stable dose of benzodiazepine.
* Have a negative alcohol breath test at screening and study start.

Exclusion Criteria:

* Have an active clinically significant unstable medical condition within 1 month (30 days) prior to screening.
* Have a history of substance dependence or substance (drug) or alcohol abuse within the 3 months before study start(nicotine and caffeine dependence are not exclusionary).
* Have a known history of neuroleptic malignant syndrome.
* Have a significant risk of suicidal or violent behavior.
* Receiving any excluded concomitant medication such as reserpine, metoclopramide, stimulants, or tetrabenazine.
* Receiving medication for the treatment of tardive dyskinesia.
* Have a positive human immunodeficiency virus antibody, (HIV-Ab), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody result at screening or have a history of positive result.
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
* Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
* Have had previous exposure with NBI-98854.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — Neurocrine Biosciences
Locations (46):
- United States (44):
  - Little Rock, Arkansas
  - Anaheim, California
  - Carson, California
  - Colton, California
  - Costa Mesa, California
  - Downey, California
  - Fountain Valley, California
  - Glendale, California
  - National City, California
  - Oceanside, California
  - Paramount, California
  - San Bernardino, California
  - San Diego, California
  - Santa Ana, California
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Lauderhill, Florida
  - Melbourne, Florida
  - Miami Springs, Florida
  - North Miami, Florida
  - Orange City, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Schaumburg, Illinois
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - St Louis, Missouri
  - Toms River, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Wards Island, New York
  - Hope Mills, North Carolina
  - Beachwood, Ohio
  - Oklahoma City, Oklahoma
  - Conshohocken, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - DeSoto, Texas
  - Irving, Texas
  - Bothell, Washington
  - Kirkland, Washington
  - Spokane, Washington
- Puerto Rico (2):
  - Caguas
  - San Juan

REFERENCES:
- [Derived] Sajatovic M, Alexopoulos GS, Burke J, Farahmand K, Siegert S. The effects of valbenazine on tardive dyskinesia in older and younger patients. Int J Geriatr Psychiatry. 2020 Jan;35(1):69-79. doi: 10.1002/gps.5218. Epub 2019 Oct 31. PMID 31617235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with a clinical diagnosis of schizophrenia or schizoaffective disorder with moderate or severe tardive dyskinesia (TD) from 35 centers in the United States and Puerto Rico. The last patient completed in October 2013.
Groups:
- Double-Blind Placebo, Then Open-Label 50mg: Double-Blind Period: Participants first received Placebo capsule (matching valbenazine capsule) once daily for 6 weeks.
  Open-Label Period: Participants received valbenazine 50mg capsule once daily for 6 weeks.
- Double-Blind 50mg, Then Open-Label 50mg: Double-Blind Period: Participants first received valbenazine 50mg capsule once daily for 6 weeks.
  Open-Label Period: Participants received valbenazine 50mg capsule once daily for 6 weeks.
- Double-Blind 100mg/50mg, Then Open-Label 50mg: Double-Blind Period: Participants first received valbenazine 100mg capsule once daily for 2 weeks, then they received valbenazine 50mg capsule once daily for 4 weeks.
  Open-Label Period: Participants received valbenazine 50mg capsule once daily for 6 weeks.
Period: Double-Blind Period (Week 0 to 6)
Arm/Group | Double-Blind Placebo, Then Open-Label 50mg | Double-Blind 50mg, Then Open-Label 50mg | Double-Blind 100mg/50mg, Then Open-Label 50mg
Started | 54 | 28 | 27
Completed | 47 | 25 | 21
Not Completed | 7 | 3 | 6
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Non-compliance | 1 | 2 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Period: Open-Label Period (Week 6 to 12)
Arm/Group | Double-Blind Placebo, Then Open-Label 50mg | Double-Blind 50mg, Then Open-Label 50mg | Double-Blind 100mg/50mg, Then Open-Label 50mg
Started | 47 | 25 | 21
Completed | 42 | 22 | 17
Not Completed | 5 | 3 | 4
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Non-compliance | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Follow-up Period (Week 12 to 16)
Arm/Group | Double-Blind Placebo, Then Open-Label 50mg | Double-Blind 50mg, Then Open-Label 50mg | Double-Blind 100mg/50mg, Then Open-Label 50mg
Started | 42 | 22 | 17
Completed | 42 | 21 | 17
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (all randomized subjects who received at least 1 dose of study drug).
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Placebo, Then Open-Label 50mg | Double-Blind 50mg, Then Open-Label 50mg | Double-Blind 100mg/50mg, Then Open-Label 50mg | Total
Number analyzed (Participants) | 54 | 28 | 27 | 109
Age, Continuous [Mean (Full Range); unit: years] | 54.5 [27 to 76] | 55.5 [42 to 72] | 55.6 [28 to 77] | 55.0 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 9 | 37
  Male | 34 | 20 | 18 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 29 | 12 | 7 | 48
  White | 23 | 15 | 19 | 57
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 1
  American Indian or Alaska Native, Black | 1 | 0 | 1 | 2
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.71 [19.2 to 44.2] | 28.85 [18.5 to 42.6] | 26.39 [14.1 to 37.8] | 28.17 [14.1 to 44.2]
Age at Schizophrenia/Schizoaffective Disorder Diagnosis [Mean (Full Range); unit: years] — Population: Date of diagnosis was not available for some subjects.
  years
    number analyzed (Participants) | 50 | 27 | 25 | 102
    (all) | 29.4 [10 to 68] | 29.7 [16 to 66] | 30.4 [17 to 66] | 29.7 [10 to 68]
Age at TD Diagnosis [Mean (Full Range); unit: years] — Population: Date of diagnosis was not available for some subjects.
  years
    number analyzed (Participants) | 49 | 26 | 22 | 97
    (all) | 46.9 [16 to 73] | 48.5 [37 to 67] | 47.5 [22 to 73] | 47.5 [16 to 73]
BPRS Total Score [Mean (Full Range); unit: units on a scale] — The Brief Psychiatric Rating Scale (BPRS) is a clinician-rated tool designed to assess change in the severity of psychopathology in patients with schizophrenia and other psychotic disorders (Overall and Gorham, 1962, 1988). The severity of each of the 18 items of the BPRS is rated on a scale of 1 (not present) to 7 (extremely severe) (total score range: 18 to 126). Higher scores represent greater symptom severity.
  units on a scale | 33.8 [20 to 48] | 32.6 [22 to 49] | 33.0 [21 to 49] | 33.3 [20 to 49]
Baseline AIMS Total Dyskinesia Score [Mean (Standard Deviation); unit: units on a scale] — The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity. Population: Baseline AIMS Total Dyskinesia Score based on the ITT analysis set.
  units on a scale
    number analyzed (Participants) | 54 | 27 | 26 | 107
    (all) | 15.3 (4.4) | 14.6 (5.9) | 14.6 (4.7) | 15.0 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score Change From Baseline at Week 6
Description: The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity. The primary efficacy endpoint was the change from baseline in the AIMS dyskinesia total score at Week 6 between the pooled NBI-98854 50+100 mg group and placebo group analyzed using the ANCOVA model (LOCF, ITT analysis set).
Time Frame: Baseline and Week 6
Population: Intent to Treat (ITT) analysis set (all subjects in the safety analysis set with an evaluable AIMS dyskinesia total score value at either Week 2 or Week 6). Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants received Placebo capsule (matching valbenazine capsule) once daily for 6 weeks.
- All Valbenazine: Includes participants who received valbenazine 50mg capsule once daily for 6 weeks and participants who received valbenazine 100mg capsule once daily for 2 weeks, then 50mg capsule once daily for 4 weeks (a total of 6 weeks).
Arm/Group | Placebo | All Valbenazine
Number analyzed (Participants) | 54 | 50
units on a scale | -2.5 (0.7) | -3.3 (0.7)
Statistical Analysis 1: Comparison: Placebo vs All Valbenazine; Test type: Other; p = 0.2966, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.3 to 0.7], Standard Error of Mean 0.8

2. Secondary Outcome: Clinical Global Impression - Global Improvement of TD (CGI-TD)
Description: Clinician's perspective of the participant's overall improvement of TD symptoms over time. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse). The ANOVA analysis of CGI-TD was conducted for the pooled NBI-98854 50+100 mg group and placebo group.
Time Frame: Week 6
Population: ITT analysis set (all subjects in the safety analysis set with an evaluable AIMS dyskinesia total score value at either Week 2 or Week 6).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Valbenazine 50mg and Valbenazine 100mg Then 50mg: Includes participants who received valbenazine 50mg capsule once daily for 6 weeks and participants who received valbenazine 100mg capsule once daily for 2 weeks, then 50mg capsule once daily for 4 weeks (a total of 6 weeks).
Arm/Group | Placebo | Valbenazine 50mg and Valbenazine 100mg Then 50mg
Number analyzed (Participants) | 54 | 50
units on a scale | 3.2 (0.1) | 3.3 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 50mg and Valbenazine 100mg Then 50mg; Test type: Other; p = 0.743, ANOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.2

3. Secondary Outcome: Clinical Global Impression - Global Improvement of TD (CGI-TD) at Week 2
Description: Clinician's perspective of the participant's overall improvement of TD symptoms over time. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse).
Time Frame: Week 2
Population: ITT analysis set (all subjects in the safety analysis set with an evaluable AIMS dyskinesia total score value at Week 2).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Valbenazine 50mg: Participants received valbenazine 50mg capsule once daily for 2 weeks.
- Valbenazine 100mg: Participants received valbenazine 100mg capsule once daily for 2 weeks.
Arm/Group | Placebo | Valbenazine 50mg | Valbenazine 100mg
Number analyzed (Participants) | 53 | 27 | 26
units on a scale | 3.6 (0.1) | 3.3 (0.2) | 3.2 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 50mg; Test type: Other; p = 0.1151, ANOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs Valbenazine 100mg; Test type: Other; p = 0.0277, ANOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.2

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Groups:
- Double-Blind 50mg: Double-Blind Period: Participants received valbenazine 50mg capsule once daily for 6 weeks.
- Double-Blind 100mg/50mg: Double-Blind Period: Participants received valbenazine 100mg capsule once daily for 2 weeks, then they received valbenazine 50mg capsule once daily for 4 weeks.
- Double-Blind Placebo: Double-Blind Period: Participants received Placebo capsule (matching valbenazine capsule) once daily for 6 weeks.
- Open-Label 50mg: Open-Label Period: Participants who completed the double-blind period entered the open-label period to receive valbenazine 50mg capsule for an additional 6 weeks of treatment.
- Follow-Up: Participants who completed the open-label period entered the 4-week follow-up period.
Arm/Group | Double-Blind 50mg | Double-Blind 100mg/50mg | Double-Blind Placebo | Open-Label 50mg | Follow-Up
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/54 | 0/93 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/27 | 1/54 | 3/93 | 0/80
Other Adverse Events (participants affected / at risk) | 4/28 | 3/27 | 2/54 | 5/93 | 1/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind 50mg (N=28) | Double-Blind 100mg/50mg (N=27) | Double-Blind Placebo (N=54) | Open-Label 50mg (N=93) | Follow-Up (N=80)
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind 50mg (N=28) | Double-Blind 100mg/50mg (N=27) | Double-Blind Placebo (N=54) | Open-Label 50mg (N=93) | Follow-Up (N=80)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.